CLINICAL TRIAL: NCT05207462
Title: A Feasibility Study of Intensive Treatment With Prolonged Exposure for Patients With Post-traumatic Stress Disorder (PTSD) in a Regular Health Care Setting
Brief Title: A Feasibility Study of Intensive Treatment With Prolonged Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Maria Bragesjo, Principal investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-06004-01
Record Dates: First submitted 2021-12-22; First posted 2022-01-26 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; prolonged exposure; intensive treatment; massed treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Prolonged exposure will be offered in a massed format with a total of nine 60 minutes sessions of imaginal exposure and processing and five 2 hour group session with psychoeducation, rationales and in vivo exposure during one treatment week followed by three individual 60 minutes sessions 2, 4 and 8 weeks afterwards.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intensive treatment with prolonged exposure (Experimental): Intensive treatment with prolonged exposure
  Interventions: Behavioral: Intensive treatment with prolonged exposure

INTERVENTIONS:
Behavioral: Intensive treatment with prolonged exposure — Intensive treatment with prolonged exposure

SUMMARY:
The primary objective with this study is to investigate the feasibility and acceptability of intensive treatment with prolonged exposure (I-PE) in regular Swedish psychiatric care. The secondary objective is to investigate preliminary effects of i-PE in terms of reducing symptoms of post-traumatic stress, depression and increase quality of life.

DETAILED DESCRIPTION:
The investigators will investigate I-PE delivered as a one-week intensive treatment consisting of nine individual sessions and five group sessions followed by three individual session two, four and eight weeks afterwards in a pilot trial. The feasibility and acceptability and preliminary effects of treatment- and assessment procedures will be evaluated using a within-group design with repeated measurements and qualitative interviews. The individual sessions will consist of imaginal exposure and processing and the group sessions of psychoeducation, rationale for treatment and in vivo exposure work. Recruitment is designed to be broadly inclusive with minimal exclusion criteria. Patients will be recruited from a psychiatric clinic specialised in PTSD in Stockholm, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for PTSD
* If taking psychotropic medication, then the dose must be stable for at least 4 weeks prior to study entry
* ≥ 18 years
* Fluent in Swedish
* Signed informed consent

Exclusion Criteria:

* Other serious comorbidity as primary concern (for example ongoing substance dependence, untreated bipolar disorder, psychotic symptoms, severe depression, high suicidal risk)
* Other ongoing trauma-focused psychological treatment
* Ongoing trauma-related threat (e.g. living with a violent spouse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Number of imaginal exposures made by the participant during the treatment period | Through treatment, up to the last session delivered eight weeks after the massed treatment week
Number of in vivo exposures made by the participant during the treatment period | Through treatment, up to up to the last session delivered eight weeks after the massed treatment week
The proportion of participants that conducts the weekly measures and further assessment points | Through study completion up to the 6 months follow up
The proportion of participants that go through the entire treatment period | Completion of treatment period, up to the last session delivered eight weeks after the massed treatment week
Adverse events related to the treatment | Through study completion, up to the 6 months follow up
  Treatment acceptability
Number of drop-outs from treatment | Completion of treatment period, up to the last session delivered eight weeks after the massed treatment week
  Treatment acceptability
Number of individuals offered the intervention but declined part of treatment | Baseline
  Treatment acceptability
Participants experience/satisfaction with treatment and assessment procedures through qualitative interviews | Completion of the massed treatment period up to post-treatment
  Qualitative interviews
Participants satisfaction with treatment, assessed by The Client Satisfaction Questionnaire (CSQ-8). | Completion of the massed treatment period (one week)
  The CSQ-8 yields a single score measuring a single dimension of overall satisfaction. An "overall score" is calculated by summing the score on each of the eight scale item. Scores range from 8 to 32, with higher values indicating higher satisfaction.

SECONDARY OUTCOMES:
Change in PTSD symptoms as assessed by the Clinician Administered PTSD Scale (CAPS-5) | Pre-treatment, 6 months follow up
  The CAPS-5 is structured interview that assesses the Diagnostic and Statistical Manual of Mental Disorders version 5 (DSM-5) criteria for PTSD (Weathers et al., 2013). Each item is rated on a severity scale ranging from 0 (Absent) to 4 (Extreme/incapacitating) and combines information about frequency and intensity for each of the 20 symptoms. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.
Change in PTSD symptoms as assessed by the PTSD Check List - DSM-5 (PCL-5) | Baseline, daily through the treatment 1 week, at the 2, 4 and 8 week sessions and the 6 months follow up.
  The PCL-5 is a 20-item self-report measure based upon the Diagnostic and Statistical Manual (DSM-5) criteria for PTSD. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.
Change in ICD-11 PTSD and complex PTSD symptoms as assessed by the International Trauma Questionnaire (ITQ). | Baseline, daily through the treatment 1 week, at the 2, 4 and 8 week sessions and the 6 months follow up.
  The ITQ includes six items measuring each PTSD symptom cluster and these items measure how bothersome each symptom has been in the past month. The ITQ also includes six items measuring each 'Disturbance in Self-Organization' (DSO) symptom in complex PTSD. These items measure how a respondent typically feels, thinks about oneself, and relates to others. The PTSD and DSO symptoms are accompanied by three items measuring associated functional impairments in the domains of social, occupation, and other important areas of life. All items are answered on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Extremely). Thus, PTSD and DSO symptom scores range from 0 to 24 and CPTSD symptom scores range from 0 to 48. Higher scores represents more PTSD and complex PTSD symptoms.
Change in depressive symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9) | Baseline, last 1 day of the treatment 1 week, at the 2, 4 and 8 week sessions and the 6 months follow up.
  The PHQ-9 is a widely used and well-validated instrument for measuring the severity of depressive symptoms. Scores are calculated based on how frequently a person experiences 9 symptoms of depression ranging from "not at all" response is scored as 0; "several days" response is 1; "more than half the days" response is 2; and "nearly every day" response is 3. Higher scores represents more depressive symptoms.
Change in quality of life measured by Euroqol, EQ-5D | Baseline, last 1 day of the treatment 1 week, at the 2, 4 and 8 week sessions and the 6 months follow up.
  Change in overall health from baseline to post treatment and follow up . EQ-5D is a standardized self-report measure of overall health status measured in terms of five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using a three-level scale: 1 having no problems, 2 having some problems and 3 having extreme problems. A higher score indicate worse severity.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bragesjö, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Traumaprogrammet, Psykiatri Sydväst, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No